CLINICAL TRIAL: NCT04322435
Title: Prevalence of Hypoglycaemia in Congenital Adrenal Insufficiency
Acronym: GLYSUR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP190910; ID RCB 2019-A02250-57 (Other: ANSM)
Record Dates: First submitted 2019-11-15; First posted 2020-03-26 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Adrenal Insufficiency, Congenital
Keywords: Congenital primary and secondary adrenal insufficiency; Cortisol deficiency; Hypoglycaemia; Children
MeSH Terms: conditions — Adrenal Insufficiency, Congenital; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adrenal insufficiency (Other): Patients followed in the paediatric endocrinology department of the Necker Hospital, with primary and secondary adrenal insufficiency, aged from 6 months to 6 years.
  Interventions: Other: Continuous blood glucose measurement; Other: Measurement of capillary blood glucose

INTERVENTIONS:
Other: Continuous blood glucose measurement — Continuous blood glucose measurement with Abbott Freestyle Pro for 14 days, repeated twice at 6 months intervals.
Other: Measurement of capillary blood glucose — Measurement of capillary blood glucose :
  * In the morning on an empty stomach, every first week of each month for 12 months.
  * In case of suspicion of hypoglycaemia (parental assessment). Abbott's Freestyle optium neo reader, used with the Accu-Chek FastClix lancing device and the Accu-Chek Performa strips.

SUMMARY:
Children with congenital primary and secondary adrenal insufficiency, who are deficient in cortisol, are at risk for hypoglycaemia, irrespective of appropriate hydrocortisone treatment, which can lead to potentially serious neurological complications. Few series are described in pediatrics. The prevalence of hypoglycaemia is probably underestimated because it is often asymptomatic and capillary blood glucose monitoring is not always performed routinely.

The objective of the study is to evaluate the prevalence of hypoglycaemia in children with adrenal insufficiency.

DETAILED DESCRIPTION:
Children with congenital primary and secondary adrenal insufficiency, who are deficient in cortisol, are at risk for hypoglycaemia, irrespective of appropriate hydrocortisone treatment, which can lead to potentially serious neurological complications. Few series are described in pediatrics. The prevalence of hypoglycaemia is underestimated because it is often asymptomatic and capillary blood glucose monitoring is not always performed routinely.

The objective of the study is to evaluate the prevalence of hypoglycaemia in children with congenital adrenal insufficiency.

The study will follow for one year children from 6 months to 6 years, with central and peripheral adrenal insufficiency.

4 study times are planned with two measurement methods:

* Continuous blood glucose measurement with Abbott Freestyle Pro for 14 days, repeated twice at 6 months intervals.
* Measurement of capillary blood glucose, in the morning on an empty stomach, every first week of each month for 12 months, with Abbott's Freestyle optium neo reader, used with the Accu-Chek FastClix lancing device and the test strips Accu-Chek performed.
* Measurement of capillary glycaemia in case of suspicion of hypoglycaemia. Measure left free according to the judgment of the parents of the necessary character or not. With Abbott's Freestyle optium neo reader, used with the Accu-Chek FastClix lancing device and the Accu-Chek performa strips.

ELIGIBILITY:
Inclusion Criteria:

* All male and female patients, followed in the Paediatric Endocrinology Department at Necker Hospital, with congenital primary and secondary adrenal insufficiency.
* Age between 6 months and 6 years.
* Included in the social security system.
* Parental consent and willingness to participate in this study: involves training and skills in the use of blood glucometers.

Exclusion Criteria:

* Patients with acquired adrenal insufficiency.
* Patients with type 1 or type 2 diabetes.
* Patients with somatotropic deficiency associated with adrenal insufficiency.
* Refusal or impossibility to perform the glycaemic measurements according to the procedure of the study.
* Not covered by the social security system.

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of hypoglycaemia | 1 year
  Number of hypoglycaemic events. Hypoglycaemia will be defined by a glucose level measured at a glucose level of less than or equal to 0.55 g /L (3 mmol /L).

SECONDARY OUTCOMES:
Duration of hypoglycaemia | 1 year
  Time in hypoglycaemia measured in minutes per day during the continuous blood glucose measurements.
Percentage of time in hypoglycaemia | 1 year
  Percentage of time in hypoglycaemia during the continuous blood glucose measurements.
Glycemic variations rate | 1 year
  Glycemic variations rate during the different measurements times: minimum rate, maximum rate, average, median. Each result will be expressed in g /L or in mmol /L. Each date will expressed by one day and for one week.
Circumstances of occurrence of hypoglycaemia | 1 year
  Circumstances in which hypoglycaemia occurred : descriptive data by parents, symptomatic or not symptomatic hypoglycaemia, descriptive signs if they are presents.
Occurrence of medical events | 1 year
  Events during the follow-up of the study: modification of treatment of hydrocortisone and fludrocortisone, re-sugaring expressed in number of sugar cubes ( by sugar cube = 20 gr of sugar) or type of sweet food given to the child, hospitalizations ( type and reason for hospitalization, cause of the decompensation).
Body Mass Index | 1 year
  Body mass divided by the square of the body height expressed in units of kg/m2 : mass in kilograms and height in meters
Systolic and Diastolic Blood Pressure | 1 year
  Expressed millimetre of mercury
Heart rate | 1 year
  Number of beats per minute
Stade tanner | 1 year
  stade tanner A1 to A5
Amount of salt consumed per day | 1 year
  Number of grams per day
Cortisol at 8 a.m. | 1 year
  microgram / deciliter
Cycle of 17-hydroxyprogesterone | 1 year
  Nanomole per liter
Adreno CorticoTropic Hormone | 1 year
  Nanogram per liter
17-hydroxyprogesterone | 1 year
  Nanomole per liter
Delta-4-Androstenedione | 1 year
  Nanomole per liter
Testosterone | 1 year
  Nanomole per liter
Ionogram | 1 year
  Nanomole per liter
Renin | 1 year
  picogram/milliliter

CONTACTS AND LOCATIONS:
Overall Officials: Dinane Samara-Boustani, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Michel Polak, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galderisi A, Kariyawasam D, Stoupa A, Quoc AN, Pinto G, Viaud M, Brabant S, Beltrand J, Polak M, Samara-Boustani D. Glucose pattern in children with classical congenital adrenal hyperplasia: evidence from continuous glucose monitoring. Eur J Endocrinol. 2023 Nov 8;189(5):K19-K24. doi: 10.1093/ejendo/lvad147. PMID 37952170